CLINICAL TRIAL: NCT01595100
Title: Anthropometric Assessment of Abdominal Obesity and Health Risk in Children and Adolescents
Acronym: Waist
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Peter T. Katzmarzyk, Associate Executive Director of Population Science, Pennington Biomedical Research Center
Other Study IDs: PBRC 29023
Record Dates: First submitted 2012-05-07; First posted 2012-05-09 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-02

CONDITIONS: Obesity
Keywords: Waist circumference; Visceral adipose tissue; Intra-abdominal fat; Pediatrics
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

SUMMARY:
Childhood obesity is a major public health issue, and the identification of children who are at increased risk of health problems due to their obesity is a priority for modern health care. Abdominal fat is considered to be the most harmful in the body, and the development of reliable landmarks and procedures for the assessment of intra-abdominal visceral adipose tissue and total body fat in children will have a major impact on 1) the early identification of children at elevated health risk, 2) the proper prioritization of health care resources, and 3) the standardization of obesity surveillance procedures within and between countries.

DETAILED DESCRIPTION:
Abdominal fat, in particular intra-abdominal visceral adipose tissue, is considered to be the most dyslipidemic and atherogenic fat depot in the human body. Intra-abdominal visceral adipose tissue and total body fat can be measured precisely and reliably in a laboratory setting using advanced imaging techniques; however, reliable clinical measurements of pediatric intra-abdominal visceral adipose tissue and total body fat are yet to be developed. Thus, the specific aims of this study are to 1) identify reliable landmarks and methodology for the measurement of pediatric waist circumference that are associated with intra-abdominal visceral adipose tissue and total body fat across the pediatric age, total body adiposity, and maturity range among African American and Caucasian children and adolescents, 2) determine if waist circumference in combination with other anthropometric indices is a better predictor of intra-abdominal visceral adipose tissue and total body fat than waist circumference alone across the pediatric age, total body adiposity, and maturation range, and 3) develop and determine the clinical utility of pediatric race-sex-specific waist circumference thresholds for the identification of elevated chronic disease risk factors across the pediatric age, total body adiposity, and maturation range. The investigators will accomplish these aims by conducting a cross-sectional study of 100 African American boys, 100 Caucasian boys, 100 African American girls, and 100 Caucasian girls 5 to 18 years of age. Waist circumference will be measured at the four common anatomic sites used in pediatric research: 1) superior border of the iliac crest, 2) midpoint between the iliac crest and the lowest rib, 3) umbilicus, and 4) minimal waist. Additional body dimensions will be obtained in order to determine the clinical utility of combining waist circumference with other measurements in predicting intra-abdominal visceral adipose tissue and total body fat, which will be assessed using advanced imaging techniques. The identification of the most appropriate waist circumference landmarks and measurement techniques is important for the clinical identification of children at elevated obesity-related health risk and for the standardization of obesity surveillance strategies within and between countries.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 5 and 18 years

Exclusion Criteria:

* Being unwilling or unable to communicate with study staff or provide informed consent
* Having a chronic medical condition or disease that is life threatening or would interfere with the measurements in this study
* Being pregnant

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Community sample from the Baton Rouge, Louisiana, metropolitan region
Sampling Method: Non-Probability Sample
Enrollment: 423 (Actual)
Dates: Start 2010-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter T Katzmarzyk, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

REFERENCES:
- [Result] Harrington DM, Staiano AE, Broyles ST, Gupta AK, Katzmarzyk PT. Waist circumference measurement site does not affect relationships with visceral adiposity and cardiometabolic risk factors in children. Pediatr Obes. 2013 Jun;8(3):199-206. doi: 10.1111/j.2047-6310.2012.00106.x. Epub 2012 Nov 21. PMID 23172858
- [Result] Broyles ST, Staiano AE, Drazba KT, Gupta AK, Sothern M, Katzmarzyk PT. Elevated C-reactive protein in children from risky neighborhoods: evidence for a stress pathway linking neighborhoods and inflammation in children. PLoS One. 2012;7(9):e45419. doi: 10.1371/journal.pone.0045419. Epub 2012 Sep 25. PMID 23049799
- [Result] Harrington DM, Staiano AE, Broyles ST, Gupta AK, Katzmarzyk PT. BMI percentiles for the identification of abdominal obesity and metabolic risk in children and adolescents: evidence in support of the CDC 95th percentile. Eur J Clin Nutr. 2013 Feb;67(2):218-22. doi: 10.1038/ejcn.2012.203. Epub 2012 Dec 12. PMID 23232587
- [Result] Barreira TV, Staiano AE, Katzmarzyk PT. Validity assessment of a portable bioimpedance scale to estimate body fat percentage in white and African-American children and adolescents. Pediatr Obes. 2013 Apr;8(2):e29-32. doi: 10.1111/j.2047-6310.2012.00122.x. Epub 2012 Dec 13. PMID 23239610
- [Result] Staiano AE, Harrington DM, Broyles ST, Gupta AK, Katzmarzyk PT. Television, adiposity, and cardiometabolic risk in children and adolescents. Am J Prev Med. 2013 Jan;44(1):40-7. doi: 10.1016/j.amepre.2012.09.049. PMID 23253648
- [Result] Staiano AE, Broyles ST, Gupta AK, Malina RM, Katzmarzyk PT. Maturity-associated variation in total and depot-specific body fat in children and adolescents. Am J Hum Biol. 2013 Jul-Aug;25(4):473-9. doi: 10.1002/ajhb.22380. Epub 2013 Apr 6. PMID 23564417
- [Result] Staiano AE, Broyles ST, Gupta AK, Katzmarzyk PT. Ethnic and sex differences in visceral, subcutaneous, and total body fat in children and adolescents. Obesity (Silver Spring). 2013 Jun;21(6):1251-5. doi: 10.1002/oby.20210. Epub 2013 May 13. PMID 23670982
- [Result] Staiano AE, Gupta AK, Katzmarzyk PT. Cardiometabolic risk factors and fat distribution in children and adolescents. J Pediatr. 2014 Mar;164(3):560-5. doi: 10.1016/j.jpeds.2013.10.064. Epub 2013 Dec 5. PMID 24315509
- [Result] Barreira TV, Broyles ST, Gupta AK, Katzmarzyk PT. Relationship of anthropometric indices to abdominal and total body fat in youth: sex and race differences. Obesity (Silver Spring). 2014 May;22(5):1345-50. doi: 10.1002/oby.20714. Epub 2014 Feb 19. PMID 24493150
- [Result] Katzmarzyk PT, Bouchard C. Where is the beef? Waist circumference is more highly correlated with BMI and total body fat than with abdominal visceral fat in children. Int J Obes (Lond). 2014 Jun;38(6):753-4. doi: 10.1038/ijo.2013.170. Epub 2013 Sep 10. No abstract available. PMID 24018751